CLINICAL TRIAL: NCT06216860
Title: The Effect of Laughter Yoga as a Nursing Intervention on Nurses' Mindfulness, Proffessional Resilience and Self-Care
Brief Title: The Effect of Laughter Yoga on Mindfulness, Proffessional Resilience and Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nuriye Yıldırım, Associate Professor, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DuzceU-SBF-NYS-01
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Laughter Yoga; Laughter Therapy; Mindfulness; Self-care
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group / Laughter yoga (Experimental): The data of the pre-intervention study will be recorded with "Personal Information Form", "Five Dimensional Mindfulness Scale" and "Skovholt Professional Resilience and Self-Care Inventory".
  The application will be done for 8 weeks, 1 day a week. Post-intervention data will be collected with "Five Dimensional Mindfulness Scale" and "Skovholt Professional Resilience and Self-Care Inventory" and "Post Laughter Yoga Evaluation Form".
  Interventions: Behavioral: Laughter Yoga
- Control group (No Intervention): The control group did not take part in the laughter yoga program. As a pre-test, the data of the study will be recorded with "Personal Information Form", "Five Dimensional Mindfulness Scale" and "Skovholt Professional Resilience and Self-Care Inventory". As the post-test, 8 weeks after the pre-test, the data of the study will be collected with the "Five Dimensional Mindfulness Scale" and "Skovholt Professional Resilience and Self-Care Inventory".

INTERVENTIONS:
Behavioral: Laughter Yoga — In Laughter Yoga Practice; each session will last approximately 30 - 45 minutes and will consist of four parts. These parts are: warm-up exercises, deep breathing exercises, childlike games and laughter exercises.
  Other Names: Interventional group
  Arms: Interventional group / Laughter yoga

SUMMARY:
The aim of this study was to evaluate the effect of laughter yoga on mindfulness, professional resilience and self-care among nurses. The hypotheses of the study suggested that laughter yoga would have an effect on mindfulness, professional resilience and self-care scores among nurses.

DETAILED DESCRIPTION:
Laughter yoga is an independent nursing intervention that includes breathing and laughter exercises. Studies have proven that laughter yoga decreases stress hormones, increases hormones such as endorphins, decreases leukocytes and provides protection against infection, accelerates circulation, increases pain tolerance and quality of life, decreases blood pressure, stress, anxiety and tension, improves mental well-being and self-esteem, improves memory and creative thinking skills, and strengthens interpersonal communication. Many of these studies have been conducted in patients, healthy adults, the elderly, nursing and university students. There are a limited number of studies in which laughter yoga was applied as an intervention in a sample of nurses. In the studies, it was determined that laughter yoga decreased cortisol hormone, fatigue levels, perceived stress, burnout levels, increased life satisfaction, attention levels and individual work performance, psychological resilience and sleep quality in nurses.

Purpose: The aim of this study was to evaluate the effect of laughter yoga on mindfulness, professional resilience and self-care among nurses.

Method:

The study is planned as an experimental research with a randomized controlled pretest-posttest control group. This study is planned to be conducted in Düzce Atatürk State Hospital between February 2024 and December 2024.

The sample size for the study was calculated using the G*Power 3.1.9.7 program. There was no article that could be taken as a reference for the scales included in this study. Therefore, taking a medium effect level (d=0.5), 5% margin of error (α=0.05), 80% power (1β=0.80) and 1:2 intervention-control group ratio, the number of people who should be included in the study according to the one-way hypothesis was found as 38 participants for the intervention group and 76 participants for the control group. Assuming drop outs, the sample size will be determined as 40 participants for the experimental group and 80 participants for the control group.

The data will be collected through "Personal Information Form", "Five Dimensional Mindfulness Scale", "Skovholt Professional Resilience and Self-Care Inventory" and "Post Laughter Yoga Evaluation Form

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Working as a nurse at Düzce Atatürk State Hospital
* Not doing laughter yoga before

Exclusion Criteria:

* Currently being in the process of any psychiatric treatment or psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Five Dimensional Mindfulness Scale Scores | Up to 8 weeks
  The Five Dimensional Mindfulness Scale developed by Baer et al. (2008), whose Turkish validity and reliability was studied by Kınay F. (2013), has 5 sub-dimensions: Acting with awareness, Identification, Observation, Not judging inner experiences, and non-reactivity to inner experiences. The scale is a 5-point Likert scale consisting of 39 questions. The internal consistency coefficient of the original scale varies between 0.75-0.91. There is no reference point in the GCBFQ. The higher the value at the end of the scale, the higher the level of mindfulness.

SECONDARY OUTCOMES:
Skovholt Professional Resilience and Self-Care Inventory Scores | up to 8 weeks
  The Turkish validity and reliability of Skovholt Professional Resilience and Self-Care Inventory developed by Skovholt (2012) was studied by Güneri et al (2017). The scale has 4 sub-dimensions: Professional wellness, Personal wellness, Professional stress and Personal stress. The scale is a 5-point Likert scale consisting of 38 questions. The total score range of the scale varies between 38 and 190, with all items being positive. High scores obtained from the scale indicate high professional resilience. The reliability coefficient of the scale was found to be 0.92.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce Üniversitesi, Düzce, Merkez, Turkey (Türkiye)